CLINICAL TRIAL: NCT01023386
Title: A Clinical Pharmacological Study to Assess the Distribution, Metabolism, and Elimination of YM155 After i.v. Infusion in Patients With Advanced Cancer
Brief Title: A Clinical Pharmacological Study of YM155 After Intravenous Infusion in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 155-CL-005; 2008-002049-21 (Other: EudraCT)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Cancer
Keywords: YM155; Mass-balance; Phase I; Pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — sepantronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YM155 — I.V.

SUMMARY:
This study investigates the pharmacokinetics of YM155, identifies the metabolic profile of YM155 and evaluates the safety and tolerability of YM155 after a 3-hour infusion in patients with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors or non-Hodgkin's lymphomas for which YM155 has the potential, based on preclinical and/or clinical data, to show efficacy, namely:

  * castrate resistant prostate cancer
  * non-small cell lung cancer
  * metastatic melanoma
  * muscle invasive bladder cancer
  * follicular lymphoma
  * diffuse large B-cell lymphoma
* Life expectancy ≥ 3 months; and Performance status (PS) ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale at baseline

Exclusion Criteria:

* Radiotherapy, major surgery, hormonal therapy, and chemotherapy within 4 weeks prior to the first dose of study medication and 6 weeks in the case of mitomycin-C or nitrosourea
* Previous therapy with YM155
* Patients with renal, hepatic or colorectal cancers
* Inadequate bone marrow, renal and/or hepatic function
* History of being treated for other malignancy within 5 years except for treated basal or squamous cell carcinoma of the skin
* Participation in any clinical study within 4 weeks prior to start of the first dose of study medication
* Known brain or leptomeningeal metastases
* Active uncontrolled systemic infection at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics, in particular the routes and extent of metabolism and excretion, of YM155 after a 3-hour infusion | Day -1 up to and including Day of discharge (Day 11)

SECONDARY OUTCOMES:
To identify the metabolic profile of YM155 | Day -1 up to and including Day of discharge (Day 11)
To evaluate the safety and tolerability of YM155 through vital signs, laboratory analysis, adverse events, physical exams, ECOG performance status and echo-cardiography | Screening (Day -21 to -2), Day -1 up to and including Day of discharge (Day 11) and end of study visit (7-14 weeks after discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Budapest, Hungary